CLINICAL TRIAL: NCT04919798
Title: Randomized, Controlled, Cross-over, First-in-man Safety and Efficacy Trial of a Novel Non-invasive Bladder Emptying Device: The NIBED Study
Brief Title: First-in-man Safety and Efficacy Trial of a Novel Non-invasive Bladder Emptying Device: The NIBED Study
Acronym: NIBED pilot
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Costs exceeding budget
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIP_NIBED_V1-8
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Urinary Retention
Keywords: Medical device; Bladder emptying; Underactive bladder; Benign prostatic obstruction; Residual urine; Non-invasive
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Underactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urinating with NIBED first, without NIBED second (Experimental): Urinating with NIBED first, without NIBED second
  Interventions: Device: Non-invasive bladder emptying device
- Urinating without NIBED first, with NIBED second (Experimental): Urinating without NIBED first, with NIBED second
  Interventions: Device: Non-invasive bladder emptying device

INTERVENTIONS:
Device: Non-invasive bladder emptying device — The NIBED is applied to the penis during urination to support bladder emptying in urinary retention patients. It is a battery-driven handheld device that is operated by the patient himself.
  Other Names: NIBED

SUMMARY:
The non-invasive bladder emptying device (NIBED) is a handheld medical device that is applied to the penis during urinating to aid bladder emptying in urinary retention patients with increased residual urine volume.

This pilot study primarily seeks to determine the safety of the NIBED. Secondary objectives are to assess the efficacy of the NIBED, which is defined as the ability of the medical device to aid or improve bladder emptying, i.e. leads to less residual urine compared to not using the NIBED.

During the intervention, the study participant will urinate with and without the NIBED. Safety variables such as penile pain, penile lesions and hematuria will be recorded. Efficacy will be assessed by measuring voided volume, residual volume, voiding time and urine flow rate.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age 18 years or older
* Sex: male
* Diagnosed with underactive bladder (UAB) (confirmed with urodynamic testing)

Exclusion Criteria:

* Acute urinary tract infection
* Patients on anti-coagulants (exception Aspirin)
* Penile pain (NPRS score >2)
* Pain during voiding (NPRS >2)
* Penile lesions (NRS score >2)
* Hematuria >2+
* Mechanical subvesical obstruction (confirmed by cystoscopy) (exception BPO)
* Transurethral resection of the prostate (TURP) less than three months before visit 2
* Penile abnormalities (Buried penis, Peyronie's disease, skin lesions)
* Asensitive bladder (no sensation of bladder fullness)
* Shy bladder
* Indwelling transurethral catheter
* Inability to understand and follow the study protocol
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Participation in another interventional clinical trial within 3 months prior to visit 2 or planned participation during the trial
* Lacking capacity for consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Penile pain | 7 days
  Assessment of penile pain (reported as numeric pain rating scale (NPRS): 0 (no pain at all) to 10 (worst imaginable pain))
Penile lesions | 7 days
  Assessment of penile lesions (visually assessed and reported as numeric rating scale (NRS): 0 (none) to 5 (exposed urethra))
Hematuria | 7 days
  Assessment of hematuria (dipstick urinalysis, scale: negative, 1+, 2+, 3+, 4+, macrohematuria (visible))
Number of patients with adverse events of special interest (AESI) | 7 days
  Number of patients with adverse events of special interest (AESI)

SECONDARY OUTCOMES:
Voided urine volume | 1 day
  Assessment of voided urine volume, measured by uroflowmeter/scale [ml]
Residual volume | 1 day
  Assessment of residual volume, measured with ultrasound bladder scanner [ml]
Voiding time | 1 day
  Assessment of voiding time, measured with clock [s]
Urine flow rate | 1 day
  Assessment of urine flow rate, measured with uroflowmeter [ml/s]

OTHER OUTCOMES:
Usability of the device | 1 day
  Assessment of usability and device acceptance, measured with a patient questionnaire (multiple choice questions and likert scale)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Kiss, Principal Investigator — Department of Urology
Locations (1):
- Bern University Hospital Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No